CLINICAL TRIAL: NCT02728869
Title: A Randomized Phase I/II Study to Evaluate Safety & Reactogenicity of Heat Stable Rotavirus Vaccine, in Healthy Adult; Followed by Evaluation of the Safety, Reactogenicity & Immunogenicity of a 3-dose Series in Infants Age 6-8 Weeks
Brief Title: Safety, Reactogenicity and Immunogenicity of Heat-stable Rotavirus Vaccine (HSRV) in Adults and Infants
Acronym: HSRV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MSD Wellcome Trust Hilleman Laboratories Pvt. Ltd. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HL/RVV/CT1/15
Record Dates: First submitted 2016-03-28; First posted 2016-04-05 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Rotavirus Gastroenteritis
MeSH Terms: interventions — Vaccines; RotaTeq

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Heat Stable Rotavirus (HSRV) Vaccine (Experimental): 25 healthy adults who will be administered a single dose of test HSRV vaccine
  Interventions: Biological: Heat Stable Rotavirus (HSRV) Vaccine
- Placebo for Heatstable Rotavirus vaccine (Placebo Comparator): 25 healthy adults who will be administered a single dose of placebo
  Interventions: Biological: Placebo for Heatstable Rotavirus vaccine
- Heat Stable Rotavirus Vaccine (Experimental): 25 healthy infants who will be administered 3-doses of test HSRV vaccine spaced at 4-week intervals
  Interventions: Biological: Heat Stable Rotavirus (HSRV) Vaccine
- RotaTeq (Active Comparator): 25 healthy infants who will be administered 3-doses of comparator Rotateq® vaccine spaced at 4-week intervals
  Interventions: Biological: RotaTeq®

INTERVENTIONS:
Biological: Heat Stable Rotavirus (HSRV) Vaccine — It is a lyophilized live attenuated pentavalent (G1-G4 and P1[8]) heat-stable rotavirus vaccine (HSRV) comprising of all the five rotavirus strains as in licensed RotaTeq® vaccine for protection against rotavirus infection
  Other Names: HSRV
  Arms: Heat Stable Rotavirus (HSRV) Vaccine; Heat Stable Rotavirus Vaccine
Biological: Placebo for Heatstable Rotavirus vaccine — It is a lyophilized formulation comprising of all the inactive ingredients as in heat stable rotavirus vaccine without any rotavirus
  Other Names: Placebo
  Arms: Placebo for Heatstable Rotavirus vaccine
Biological: RotaTeq® — It is a pentavalent human-bovine (WC3) reassortant live-attenuated, oral vaccine developed by Merck Research Co., West Point, Pennsylvania, USA. This vaccine contains five live reassortant rotaviruses. Four reassortant rotaviruses express the VP7 protein (G1, G2, G3, or G4) from the human rotavirus parent strain and the attachment protein (P7[5]) from bovine rotavirus parent strain WC3. The fifth reassortant virus expresses the attachment protein (P1A[8]) from the human rotavirus parent strain and the outer capsid protein G6 from the bovine rotavirus parent strain.
  Other Names: Active Comparator
  Arms: RotaTeq

SUMMARY:
Rotaviruses are the leading cause of severe, dehydrating diarrhoea and related deaths in children aged less than 5 years worldwide and are reported to infect nearly every child by the age of 5 years. About 90% of all rotavirus-associated fatalities occur in low income countries in Africa and Asia and are related to poor health care. In view of high global RVGE burden, the World Health Organization (WHO) on 5th June 2009, recommended the inclusion of rotavirus vaccine in all the national immunization programs.

Currently available rotavirus vaccines, RotaTeq® and Rotarix®, are WHO prequalified vaccines which are stable for recommended duration at storage temperature between 2-8 °C. However, if these vaccine are exposed to temperatures above 30 °C, the vaccine has to be discarded due to lost potency. It is very difficult to maintain the cold chain required to conserve the vaccine potency particularly in developing and low income countries, resulting in large amount of vaccine being wasted and in worst case scenario, endangering the lives of potential recipients. The WHO estimates that nearly half of freeze-dried and quarter of liquid vaccines are wasted each year. One of the biggest contributors to this wastage is disruption of the cold chain systems.

Hilleman Labs new Rotavirus vaccine is a lyophilized heat stable rotavirus vaccine comprising of five live attenuated reassortant rotaviruses similar to RotaTeq®. The new heat stable rotavirus vaccine (HSRV) formulation offers a stability profile of 9 months at 45 °C and 12 months at 37 °C. This new heat stable formulation (HSRV) could be transported in non-refrigerated supply chain significantly reducing the cost and complications associated with transporting vaccine to remote corners of the developing world. Heat-stable rotavirus vaccine (HSRV) has a potential to sustain high temperatures frequently encountered in regions where majority of rotavirus burden exists and has potential to partially or completely eliminate cold chain dependence.

The current study has been designed to test for the first time in humans, the safety and tolerability of the new heat stable rotavirus vaccine (HSRV) in adults; followed by safety and immunogenicity in infants of age 6-8 weeks, as compared to the licensed RotaTeq® vaccine.

DETAILED DESCRIPTION:
Rotaviruses are the leading cause of severe, dehydrating diarrhea and related deaths in children aged less than 5 years worldwide and are reported to infect nearly every child by the age of 5 years. About 90% of all rotavirus-associated fatalities occur in low income countries in Africa and Asia and are related to poor health care. In most low income countries in Asia and Africa, rotavirus epidemiology is characterized by one or more periods of relatively intense rotavirus circulation against a background of year-round transmission, whereas in high income countries with temperate climates a distinct winter seasonality is typically observed. In 2008, WHO estimated approximately 453,000 (420,000-494,000) rotavirus gastroenteritis (RVGE) associated child deaths worldwide. These fatalities accounted for about 5% of all child deaths with a cause-specific mortality rate of 86 deaths per 100,000 population aged less than 5 years. In view of high global RVGE burden, the World Health Organization (WHO) on 5th June 2009, recommended the inclusion of rotavirus vaccine in all the national immunization programs.

As in other Asian countries, Rotavirus infection is a significant cause of illness and hospitalizations in Bangladesh with approximately 2.4 million cases being reported every year and nearly two-thirds of all diarrhea-related hospitalizations in children under age 5. While progress has been made in reducing diarrhea-related deaths among children, it is still one of the leading causes of illness among children under 5 in Bangladesh. About half of all rotavirus hospitalizations were among infants age 6-11 months, Rotavirus vaccines could have a powerful public health impact if introduced into Bangladesh's national immunization program.

The basis for developing a rotavirus vaccine rested on the observation that wild-type rotavirus infection immunized children against subsequent disease. The immunity from wild-type infection does not prevent all subsequent infections; however, it provides nearly complete protection against severe disease and substantial protection against mild disease. The five most prevalent rotavirus genotype/serotype combinations are G1P1A[8], G2P1B[4], G3P1A[8], G4P1A[8], and G9P1A[8].

Currently, RotaTeq® and Rotarix® are the two WHO prequalified vaccines which are stable for recommended duration at storage temperature between 2-8 °C. Studies indicate that if these currently available vaccine, for example RotaTeq®, is inadvertently exposed or stored at temperatures above 8 °C, the potency is maintained for the maximum exposure of 48 hours at 9 °C to 25 °C or for a bare 12 hours at 26 °C to 30 °C. However, if RotaTeq® vaccine is exposed to temperatures above 30 °C, the vaccine has to be discarded due to lost potency. There is limited data to suggest that if the vaccine is inadvertently exposed to temperatures below 0 °C, the potency of the vaccine is maintained. Another, currently available freeze dried vaccine i.e. Rotarix® vaccine exhibits stability with a shelf life of 36 months at 2 °C to 8 °C.

Hence these vaccines do not possess enough thermostability profile suitable for storage outside cold chain for any meaningful amount of time and needs to be stored and transported under refrigeration. It is very difficult to maintain the cold chain required to conserve the vaccine potency particularly in developing and low income countries, resulting in large amount of vaccine being wasted and in worst case scenario, not providing protection against rotavirus infection to potential recipients. Many other existing vaccines do exhibit some degree of thermostability, however, the existing licensed vaccines possess shorter period of thermostability (e.g. VVM 7 or VVM 14) which fails to address the issues in developing countries especially in region of extreme climatic conditions, reaching up to 40 °C.

Heat Stable Rotavirus Vaccine is a lyophilized heat stable rotavirus vaccine comprising of five live reassortant rotaviruses in RotaTeq®. The parent strains of the reassortants were isolated from human and bovine hosts. Four reassortant rotaviruses express one of the outer capsid proteins (G1, G2, G3, or G4) from the human rotavirus parent strain and the attachment protein (P7) from the bovine rotavirus parent strain. The fifth reassortant virus expresses the attachment protein, P1A (genotype P[8]), referred to as P1[8], from the human rotavirus parent strain and the outer capsid protein G6 from the bovine rotavirus parent strain. These reassortants were suspended in stabilizer solution which was then lyophilized to obtain thermostable cake. This lyophilized cake will be reconstituted using a reconstitution buffer. There are no preservatives or thimerosal present in the vaccine. The new heat stable rotavirus vaccine (HSRV) formulation offers higher titer value even at extreme temperature conditions up to 45 °C for prolonged periods of time. This new heat stable formulation (HSRV) could be transported in non-refrigerated supply chain significantly reducing the cost and complications associated with transporting vaccine to remote corners of the developing world. The bulk of reassortants virus have been procured directly from Merck and Co., USA, currently licensed in USA and many countries as liquid formulation RotaTeq®, offering an easier regulatory path for new heat-stable rotavirus vaccine licensure & WHO prequalification. Heat-stable rotavirus vaccine (HSRV) has a potential to sustain high temperatures frequently encountered in regions where majority of rotavirus burden exists and has potential to partially or completely eliminate cold chain dependence.

The aim of the current study is to assess the safety and reactogenicity of a single dose of Hilleman Labs.' oral live attenuated HSRV vaccine in healthy adults aged 18 years to 45 years followed by safety & immunogenicity evaluation in infant population 6-8 weeks of age. In current study, adult subjects will either receive a single dose of oral live attenuated HSRV vaccine or placebo at Day 0. There will be a safety follow-up for all subjects for a period of 14 days after vaccination. The investigators intend to establish the safety of HSRV in healthy adults prior to testing in infant population. Acceptable safety data from the adult cohort will allow enrolment of subjects in the infant cohort, after approval from study DSMB.

ELIGIBILITY:
Inclusion Criteria:

Healthy Adults:

1. Healthy adult subjects of either sex, between 18 to 45 years of age;
2. No apparent signs or symptoms of ill health;
3. Subjects properly informed about the study and having signed the informed consent form (ICF). In case of subjects' inability to read or write, having had the ICF explained to them in the presence of a study independent witness and the witness having signed the ICF;
4. Subjects' availability for the entire period of the study and reachability by study staff for post vaccination follow-up.

Healthy Infants:

1. Healthy infants of either sex, 6-8 weeks of age at the time of enrollment;
2. Born after a gestational period of 36-42 weeks with birth weight ≥ 2kg;
3. Father, mother or other legally authorized representative (guardian) properly informed about the study and having signed the informed consent form (ICF). In case of father's, mother's or other legally acceptable representative's (guardian) inability to read or write, having had the ICF explained to them in the presence of a study independent witness and the witness having signed the ICF;
4. Infant/Parents' or guardian's availability for the entire period of the study and reachability by study staff for post-vaccination follow-up.

Exclusion Criteria:

Healthy adults:

1. Known or suspected impairment of immunological function; and known immunosuppressed family members/household contacts
2. Known hypersensitivity to any component of the rotavirus vaccine;
3. Fever, with axillary temperature ≥38.1 oC (≥100.5 oF) as measured by study staff;
4. History of chronic diarrhea;
5. Clinical evidence of active gastrointestinal illness;
6. Receipt of any IM, oral, or IV corticosteroid treatment in the past 30 days;
7. Subjects' suspected to be HIV, HBV or HCV positive from the available clinical history;
8. Any subject who cannot be adequately followed for safety assessment;
9. Any conditions which, in the opinion of the investigator, might interfere with the evaluation of the study objectives;
10. Subject's inability to maintain diary card;
11. Participation in another clinical trial investigating a vaccine, drug, medical device or medicinal procedure in the 4 weeks preceding the current vaccination trial;
12. Planned participation in another clinical trial during the present trial period;
13. Subjects identified as employees of the investigator or study center, with direct involvement in the proposed study or studies under the direction of that investigator or study center as well as children, adopted or natural, of the employees or Investigator.

Healthy Infants:

1. History of congenital abdominal disorders, intussusception, or abdominal surgery;
2. Infants exhibiting signs of severe malnutrition or Known or suspected impairment of immunological function(s) in subject or his/her immediate family;
3. Developmental delay or neurological disorder;
4. Known hypersensitivity to any component of the rotavirus vaccine;
5. Prior receipt of any rotavirus vaccine;
6. Prior receipt of any dose of Diphtheria, Tetanus, Pertussis, Hepatitis B, Hib or polio virus containing vaccine(s). Birth dose of Hepatitis B and Oral Polio Vaccine is allowed to be administered to the infants as per the local immunization practices. Oral Polio Vaccines administered as a part of the National Pulse Polio Program are allowed to be administered to the infants.
7. Fever, with axillary temperature ≥38.1 oC (≥100.5 oF) as measured by study staff.
8. History of known rotavirus disease, chronic diarrhea, or failure to thrive;
9. Clinical evidence of active gastrointestinal illness including ongoing diarrheal episode (infants with GERD can participate in the study so long as this condition is well controlled with or without medication);
10. Receipt of any IM, oral, or IV corticosteroid treatment in the past 30 days (infants on inhaled steroids may be permitted to participate in the study);
11. Infants residing in a household with an immuno-compromised person (e.g., individuals with a congenital immunodeficiency, HIV infection, leukemia, lymphoma, Hodgkin's disease, multiple myeloma, generalized malignancy, chronic renal failure, nephritic syndrome, organ or bone marrow transplantation, or those receiving immunosuppressive chemotherapy including long-term systemic corticosteroids);
12. Infants already laboratory-confirmed or suspected to be HIV, HBV or HCV positive from the available clinical history or born to mothers known to be HIV, HBV or HCV positive (no specific screening for the purpose of the study would be carried out);
13. Prior receipt of a blood transfusion or blood products, including immunoglobulins, in the past 4 weeks which might interfere with the assessment of the immune response;
14. Any infants who cannot be adequately followed for safety assessment by a home visit;
15. Any conditions which, in the opinion of the investigator, might interfere with the evaluation of the study objectives;
16. Parent/s or guardian of infant unable to maintain symptom diary;
17. Participation in another clinical trial investigating a vaccine, drug, medical device or medicinal procedure in the 4 weeks preceding the current vaccination trial;
18. Planned participation in another clinical trial during the present trial period;
19. Parents/ Guardians/ Legally Authorized Representatives identified as employees of the investigator or study center, with direct involvement in the proposed study or studies under the direction of that investigator or study center as well as children, adopted or natural, of the employees or Investigator.

    -

Ages: 6 Weeks to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Any adverse event in adult cohort | Up to two weeks after single dose of vaccine or placebo
Serious adverse events in adult cohort | Up to two weeks after single dose of vaccine or placebo
Any adverse event in infant cohort | Up to one month after 3 doses of vaccine or active control
Serious adverse events in infant cohort | Up to one month after 3 doses of vaccine or active control

SECONDARY OUTCOMES:
Anti-Rotavirus IgA sero-response rate in infant cohort | One month after third dose of vaccine or active control
  Serum IgA response rates, defined as the proportion of subjects with positive three-fold sero-response (i.e. a threefold rise in serum IgA anti-rotavirus antibody titres from baseline) 28 days after administration of third dose of investigational and comparator vaccine.
Viral shedding after single dose of vaccine or placebo in adults | Up to 7 days after single dose of vaccine or placebo
Viral shedding in infants after each dose of vaccine or active control in infants | Up to 7 days after each dose of vaccine

CONTACTS AND LOCATIONS:
Overall Officials: K Zaman, MBBS, PhD, Principal Investigator — International Center for Diarrheal Disease Research, Bangladesh
Locations (1):
- Icddr,B, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided
Will disclose de-identified data of all subject after completion of study

REFERENCES:
- [Derived] Kanchan V, Zaman K, Aziz AB, Zaman SF, Zaman F, Haque W, Khanam M, Karim MM, Kale S, Ali SK, Goveia MG, Kaplan SS, Gill D, Khan WA, Yunus M, Singh A, Clemens JD. A randomized Phase I/II study to evaluate safety and reactogenicity of a heat-stable rotavirus vaccine in healthy adults followed by evaluation of the safety, reactogenicity, and immunogenicity in infants. Hum Vaccin Immunother. 2020 Mar 3;16(3):693-702. doi: 10.1080/21645515.2019.1664239. Epub 2019 Oct 29. PMID 31526218